CLINICAL TRIAL: NCT02006095
Title: Neuroimaging Correlates of Memory Decline Following Carotid Interventions
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: R21NS081416-01 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2013-12-09 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stenting; carotid endarterectomy; magnetic resonance imaging (MRI); neuropsychological testing; microemboli
MeSH Terms: conditions — Carotid Stenosis | interventions — Magnetic Resonance Spectroscopy; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neuroimaging Correlates
  Interventions: Other: Magnetic resonance imaging; Behavioral: Neuropsychological testing

INTERVENTIONS:
Other: Magnetic resonance imaging — arterial spin labeling, diffusion tensor imaging, and diffusion weighted imaging sequences will be used
Behavioral: Neuropsychological testing

SUMMARY:
Carotid revascularization can significantly reduce the risk of stroke in patients with severe carotid stenosis; however, it has been associated with cognitive decline in 25% of the older adults who undergo the procedure. Characterizing risk factors for cognitive decline following carotid interventions and individualizing treatment strategy based on those risks can minimize procedure-associated cognitive dysfunction. Neuroimaging techniques that characterize white matter integrity and regional hypoperfusion have the potential to provide sensitive brain structure indicators that may be associated with memory decline following revascularization procedures. In this protocol, we hope to determine how cerebral blood flow and baseline white matter abnormality in the vulnerable region modify the frequency and cognitive effect of microembolization following carotid revascularization procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female >40 yrs of age.
* Patient has occlusive extracranial carotid stenosis (≥70%)
* Patient is scheduled to undergo a carotid revascularization procedure
* Patient agrees to voluntarily participate in the study and signs an informed consent.
* Patient agrees to be available for follow-up and is able to participate in all study testing procedures.
* Patient has sufficient visual and auditory acuity for cognitive testing.

Exclusion Criteria:

* Patient is unable to safely and comfortably undergo MR imaging procedures (e.g., claustrophobia, implanted medical devices that are MRI incompatible such as pacemaker, defibrillator, neural stimulator etc)
* Patient has an untreated or unsuccessfully controlled psychiatric disease (schizophrenia, bipolar disorder).
* Patient has prominent suicidal or homicidal ideation.
* Patient has acute illness or unstable chronic illness (e.g. uncontrolled hypertension, hepatic encephalopathy, portal hypertension, ascites, and esophageal varices, pancreatitis).
* Patient with a history of neurological (e.g., multiple sclerosis, seizure disorder, Parkinson's disease) or systemic illness affecting central nervous system function.
* Patient has prior closed head injury with ≥24 hours of amnesia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid intervention
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Brain MRI scans | 6 months following the procedure
  White matter abnormality and perfusion in correlation with microembolization and cognitive change

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhou, MD, Principal Investigator — Palo Alto Veterans Affairs/Stanford University
Locations (1):
- Palo Alto Veterans Affairs, Palo Alto, California, United States